CLINICAL TRIAL: NCT03369795
Title: A Randomized Double Blind Parallel Trial Administering Methotrexate vs Placebo as add-on to Antipsychotics in Patients With Schizophrenia or Schizoaffecive Disorder
Brief Title: Add-on Methotrexate for the Treatment of Schizophrenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-17-3512-MW-CTIL
Record Dates: First submitted 2017-12-03; First posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Schizophrenia
Keywords: methotrexate; add-on; schizophrenia; schizoaffective
MeSH Terms: conditions — Schizophrenia | interventions — Methotrexate; Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Drug (Experimental): Methotrexate 10mg
  Interventions: Drug: Methotrexate
- Placebo (Placebo Comparator): Pills equivalent to other study arm (10 mg)
  Interventions: Other: Placebo Arm

INTERVENTIONS:
Drug: Methotrexate — Methotrexate 10mg once a week will be given for the first two weeks of the trial, followed by an increase in dose to 15mg or equivalent placebo once a week until week 16.
  Other Names: Study Drug
  Arms: Study Drug
Other: Placebo Arm — Pills equivalent to the study drug arm (10mg) will be given once a week for the first two weeks of the trial, followed by an increase in dose to 15mg of equivalent placebo once a week until week 16.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
A recent double-blind placebo-controlled study has tested the effect of methotrexate as an add-on treatment for patients with schizophrenia or schizoaffective disorder, administering 10 mg of methotrexate or placebo once a week for a period of three months to 72 patients (Chaudry, Husain et al. 2015). Results showed improvement both in positive symptoms, as measured by the Positive symptoms subscale of the Positive and Negative Syndrome Scale (PANSS), and in total PANSS scores.

The objective of this study is to replicate Chaudry et al.'s study. This proposed study will randomize schizophrenia or schizoaffective disorder patients to methotrexate or placebo for a period of four months.

The study will enroll patients with a DSM-IV-TR diagnosis of schizophrenia or schizoaffective disorder confirmed by the Modified Structured Clinical Interview for Diagnosis (SCID). In order to be eligible to enter the study, the patient must have a score of 4 (moderately ill) or greater on the Clinical Global Impression - Severity (CGI-S) scale. In addition, inclusion criteria reflect patients with moderate or more severity on positive symptoms, hence having a score of 4 (moderate) or above on two of the following four PANSS items: delusions, hallucinatory behaviors, conceptual disorganization or suspiciousness/ persecution. Patients receiving more than one anti-psychotic or depot antipsychotic will be allowed to participate, and patients receiving anti-cholinergic agents, beta-blockers, anti-depressants, mood-stabilizers, sedatives, and anti-anxiety agents will be allowed in the study. Because the clinical status of patients sometimes improves in the days following admission to the hospital, newly hospitalized patients will have their baseline visit 3 days or more after being hospitalized.

DETAILED DESCRIPTION:
OBJECTIVES The objective of the study is to evaluate the efficacy of Methotrexate compared to placebo, as add-on to anti-psychotics in the treatment of patients with schizophrenia or schizoaffective disorder.

ENDPOINTS Primary outcome measure: PANSS positive score at the end of the trial. Secondary outcome measures: PANSS total, negative and general psychopathology scales, Clinical Global Impression Scale-Severity (CGI-S) and Global Impression Scale-Improvement (CGI-I), Social Functioning Scale Assessment (PSP) and rates of drop outs before the end of the trial.

DESIGN Randomized, add-on to anti-psychotics, double blind, placebo-controlled trial.

ASSESSMENTS

* Positive and Negative Syndrome Scale (PANSS). PANSS is a 30-item rating scale widely used in assessment of medication effects in schizophrenia.
* Clinical Global Impression-Severity (CGI-S) and Clinical Global Impression-Improvement (CGI-I). CGI-S and CGI-I will be used to assess severity of the illness and global improvement.
* The Udvalg for Kliniske Undersogelser (UKU) Side Effect Rating Scale: will be used to assess commonly occurring side effects caused by anti-psychotics.
* The methotrexate toxicity checklist includes rash, oral ulceration, nausea and vomiting, diarrhea, new or increasing dyspnea, new or increasing dry cough, severe sore throat, and abnormal bruising.
* The Personal and Social Performance (PSP) scale will be used to assess social functioning.

PROCEDURE At the screening visit informed consent will be obtained, inclusion and exclusion criteria will be examined, and demographic information will be collected. The PANSS, CGI-S and SCID assessment will be administered, a physical examination will be done, psychiatric and medical history obtained, and blood samples for chemistry and CBC, and urine samples for urinalysis will be taken. Patients will liver function levels higher than normal will be excluded. Females of child-bearing potential will be tested for pregnancy. Patients will be screened for HIV, Hepatitis B and C.

At the baseline visit, The PANSS, CGI-S, UKU, and PSP will be administered. Patients will be randomized to start study medication: Methotrexate 10 mg/week or equivalent dose of placebo will be administered to patients. Medication dose will start at 10mg for the first two weeks and will then be increased to 15 mg. Patients will also be instructed to take 5 mg/day of folic acid for 6 days/week in order to avoid vitamin deficiencies due to the methotrexate use. In order to monitor potential side-effects, blood tests for CBC and SMA will be taken at screening, week 2, week 4, week 8, week 12, and week 16 (EOS).

Subjects will be assessed at clinic visits according to timelines described above. Additionally, during the weeks in which patients will not come for clinic visits, they will have phone visits in order to monitor medication adherence and adverse events. Throughout all the visits between baseline and end of study, patients will be checked for methotrexate toxicity using the methotrexate toxicity checklist which inquires for includes rash, oral ulceration, nausea and vomiting, diarrhea, new or increasing dyspnea, new or increasing dry cough, severe sore throat, and abnormal bruising.

A final, End-of-Study, clinical evaluation will occur on Week 16, or at the time of early discontinuation from the study, and will include a physical examination; vital signs; rating of the PANSS, CGI-S, CGI-I, UKU, PSP, review of adverse events, methotrexate toxicity checklist and concomitant medications. Blood samples will be taken for SMA, CBC, and urine samples for urinalysis. Females of child-bearing potential will be tested for pregnancy, and a blood sample for medication levels will be taken.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-35 years of age, inclusive
2. Females who are abstinent or practicing an established method of birth control (oral contraceptive tablets, hormonal implant device, hormone patch, injectable contraceptive, intrauterine device [IUD]).
3. Willing and able to provide informed consent, after the nature of the study has been fully explained.
4. Current DSM-IV-TR diagnosis of schizophrenia or schizoaffective disorder as confirmed by modified SCID.
5. Within the first five years of diagnosis.
6. Positive symptoms: 4 (moderate) or above on CGI-S and a score of 4 (moderate) or above on two of the following four PANSS items: delusions, hallucinatory behaviors, conceptual disorganization or suspiciousness/ persecution.
7. Receiving only one anti-psychotic within PORT dosages
8. Inpatients or outpatients. Inpatients will be randomized 3 days or more after admission

Exclusion Criteria:

1. Unwilling or unable, in the opinion of the Investigator, to comply with study instructions
2. Evidence of significant liver disease. Patients with LFT above normal will be excluded.
3. Pregnant or breast-feeding
4. Unstable medical disease (malignancy, poorly controlled diabetes, active ischemic cardiac disease, or cardiomyopathy, serious pulmonary disease, COPD and other chronic lungs diseases, serious hematological disorder, kidney disease, impaired liver functioning)
5. At significant risk of committing suicide, or in the opinion of the Investigator, currently is at imminent risk of suicide or harming others.
6. Patients with a current DSM-IV substance or alcohol abuse. Patients with a history of and/or current recreational use of cannabinoids or alcohol, and/or patients who smoke cigarettes can be included.
7. Concurrent delirium, mental retardation, drug-induced psychosis, or history of clinically significant brain trauma documented by CT or MRI.
8. Lactose intolerance
9. Immune system disorder or serious infection
10. Patients taking Clozapine

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-15 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
PANSS (Positive and Negative Syndrome Scale) Positive Subscale Score at the end of the trial | Changes throughout 16 weeks
  The positive score subscale has a minimum score of 7 and a maximum score of 49, 7 showing no symptomatology, and 49 showing very severe symptomatology

SECONDARY OUTCOMES:
PANSS (Positive and Negative Syndrome Scale) Total score at the end of the trial | Changes throughout 16 weeks
  The PANSS scale has a minimum score of 30 and a maximum score of 210, 30 showing no symptomatology, and 210 showing very severe symptomatology
PANSS (Positive and Negative Syndrome Scale) Negative Susbcale Score at the end of the trial | Changes throughout 16 weeks
  The negative score subscale has a minimum score of 7 and a maximum score of 49, 7 showing no symptomatology, and 49 showing very severe symptomatology
PANSS (Positive and Negative Syndrome Scale) General Psychopathology Subscale Score at the end of the trial | Changes throughout 16 weeks
  The general psychopathology subscale score has a minimum score of 16 and a maximum score of 112, 16 showing no symptomatology, and 112 showing very severe symptomatology
Clinical Global Impression Scale- Severity (CGI-S) at the end of the trial | Changes throughout 16 weeks
  This is a clinical scale with a minimum score of 1 (not ill) and a maximum score of 7 (among the most extremely ill patients)
Clinical Global Impression Scale- Improvement (CGI-I) at the end of the trial | Changes throughout 16 weeks
  This is a clinical scale with a minimum score of 1 (very much improved) and a maximum score of 7 (very much worse)
Social Functioning Scale Assessment (PSP) at the end of the trial | Changes throughout 16 weeks
  This is a social functioning scale with a minimum score of 1 (no functioning) and a maximum score of 100 (excellent functioning)
Rates of drop outs before the end of the trial | Rates throughout 16 weeks
  The number of drop outs from the study will be analysed at the end of the study.